CLINICAL TRIAL: NCT00620022
Title: A Phase III Randomized, Double-blind, Placebo-controlled, 2-period Crossover, Multicenter Study to Assess the Effect of Indacaterol (300 μg o.d.) on Exercise Endurance in Patients With Moderate to Severe Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: The Effect of Indacaterol on Exercise Endurance in Patients With Moderate to Severe Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CQAB149B2311
Record Dates: First submitted 2008-02-08; First posted 2008-02-21 (Estimated); Results first posted 2011-08-17 (Estimated); Last update posted 2011-08-17 (Estimated); Status verified 2011-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: indacaterol; chronic obstructive pulmonary disease; exercise endurance; moderate to severe chronic obstructive pulmonary disease; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — indacaterol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Indacaterol 300 μg followed by placebo (Experimental): Patients first received indacaterol 300 μg delivered via a single dose dry powder inhaler (SDDPI) once daily (od) in the morning for 3 weeks. After a 3-week washout period, patients received placebo delivered od via a SDDPI in the morning for 3 weeks. Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. The short-acting β2-agonist salbutamol/albuterol was available for rescue use throughout the study.
  Interventions: Drug: Indacaterol 300 μg; Drug: Placebo
- Placebo followed by indacaterol 300 μg (Experimental): Patients first received placebo delivered via a single dose dry powder inhaler (SDDPI) once daily (od) in the morning for 3 weeks. After a 3-week washout period, patients received indacaterol 300 μg delivered od via a SDDPI in the morning for 3 weeks. Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. The short-acting β2-agonist salbutamol/albuterol was available for rescue use throughout the study.
  Interventions: Drug: Indacaterol 300 μg; Drug: Placebo

INTERVENTIONS:
Drug: Indacaterol 300 μg — Indacaterol was supplied in powder filled capsules together with a single dose dry powder inhaler (SDDPI) device.
Drug: Placebo — Placebo was supplied in powder filled capsules together with a single dose dry powder inhaler (SDDPI) device.

SUMMARY:
This study compared the effect of indacaterol (300 μg once daily [od]) on exercise endurance with that of placebo in patients with moderate to severe chronic obstructive pulmonary disease.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults aged ≥ 40 years, who have signed an informed consent form prior to initiation of any study-related procedure.
* Co-operative outpatients with a diagnosis of moderate to severe chronic obstructive pulmonary disease (COPD), as classified by the GOLD Guidelines (2006), and:

  * Smoking history of at least 20 pack years.
  * Post-bronchodilator forced expiratory volume in 1 second (FEV1) < 80% and ≥ 30% of the predicted normal value.
  * Post-bronchodilator FEV1/forced vital capacity (FVC) < 70%.

Exclusion Criteria:

* Pregnant or nursing (lactating) women.
* Women of child-bearing potential.
* Patients who have been hospitalized for a COPD exacerbation in the 6 weeks prior to screening or during the run-in period.
* Patients requiring oxygen therapy or who experience oxygen desaturation to < 80% during cycle exercise on room air.
* Patients with a Wmax value < 20 W (as determined by the incremental cycle endurance test) at screening.
* Patients who have had a respiratory tract infection within 6 weeks prior to screening.
* Patients with contra-indications of cardiopulmonary exercise testing.
* Patients with concomitant pulmonary disease.
* Patients with a history (up to and including the screening visit) of asthma.
* Patients with diabetes Type I or uncontrolled diabetes Type II.
* Any patient with lung cancer or a history of lung cancer.
* Any patient with active cancer or a history of cancer with less than 5 years disease free survival time.
* Patients with a history of long QT syndrome or whose QTc interval (Bazett's) measured at the collection of informed consent visit (Visit 1) or randomization is prolonged.
* Patients who have been vaccinated with live attenuated vaccines within 30 days prior to screening or during the run-in period.
* Patients unable to successfully use a dry powder inhaler device, metered dose inhaler (MDI), or perform spirometry measurements.

Other protocol-defined inclusion/exclusion criteria applied to the study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2008-04; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharma, Study Chair — Novartis Pharmaceuticals
Locations (20):
- United States (2):
  - Novartis Investigator Site, Torrance, California
  - Novartis Investigator Site, Lebanon, New Hampshire
- Belgium (4):
  - Novartis Investigator Site, Brussels
  - Novartis Investigator Site, Gembloux
  - Novartis Investigator Site, Jette
  - Novartis Investigator Site, Liège
- Canada (2):
  - Novartis Investigator Site, Edmonton
  - Novartis Investigator Site, Kingston
- Denmark (4):
  - Novartis Investigator Site, Aarhus
  - Novartis Investigative Site, Hellerup
  - Novartis Investigator Site, Hvidovre
  - Novartis Investigative site, Odense
- Italy (3):
  - Novartis Investigator Site, Genova
  - Novartis Investigator Site, Pisa
  - Novartis Investigator Site, Verona
- Spain (5):
  - Novartis Investigator Site, Alicante
  - Novartis Investigator Site, Barcelona
  - Novartis Investigative Site, Madrid
  - Novartis Investigative site, Seville
  - Novartis Investigator Site, Zaragoza

REFERENCES:
- [Derived] O'Donnell DE, Casaburi R, Vincken W, Puente-Maestu L, Swales J, Lawrence D, Kramer B; INABLE 1 study group. Effect of indacaterol on exercise endurance and lung hyperinflation in COPD. Respir Med. 2011 Jul;105(7):1030-6. doi: 10.1016/j.rmed.2011.03.014. Epub 2011 Apr 16. PMID 21498063

RESULTS

PARTICIPANT FLOW:
Period: Treatment Period 1
Arm/Group | Indacaterol 300 μg Followed by Placebo | Placebo Followed by Indacaterol 300 μg
Started | 46 | 43 (Of 44 randomized patients, 1 patient discontinued before receiving any study treatment.)
Completed | 41 | 37
Not Completed | 5 | 6
Not completed — Adverse Event | 4 | 6
Not completed — Subject withdrew consent | 1 | 0
Period: Treatment Period 2
Arm/Group | Indacaterol 300 μg Followed by Placebo | Placebo Followed by Indacaterol 300 μg
Started | 41 | 37
Completed | 39 | 35
Not Completed | 2 | 2
Not completed — Adverse Event | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: The entire study population includes the group of patients who received indacaterol 300 μg in the first treatment period followed by placebo in the second treatment period and the group of patients who received placebo in the first treatment period followed by indacaterol 300 μg in the second treatment period. Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. The short-acting β2-agonist salbutamol/albuterol was available for rescue use throughout the study.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 89
Age Continuous [Mean (Standard Deviation); unit: years] | 62.8 (8.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 62

OUTCOME MEASURES:

1. Primary Outcome: Exercise Duration Time Assessed by Constant-load Cycle Ergometry at the End of Each Treatment Period
Description: At the end of each 3 week treatment period, patients completed constant-load cycle ergometry testing at a work-rate of 75% of the Wmax determined at Screening. This work-rate was maintained until symptom limitation caused the patient to stop exercising. The time from the start of loaded pedaling until the patient stopped exercising was recorded.
Time Frame: End of each 3 week treatment period (last day of Weeks 3 and 9)
Population: Modified intent-to-treat (modified ITT) population: All randomized patients who received at least 1 dose of study drug. The number of patients analyzed for each treatment group was the number with non-missing values for the dependent and independent variables in the mixed model.
Measure: Least Squares Mean (Standard Error); unit: Seconds
Groups:
- Indacaterol 300 μg: Patients received indacaterol 300 μg delivered via a single dose dry powder inhaler (SDDPI) once daily (od) in the morning for 3 weeks. Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. The short-acting β2-agonist salbutamol/albuterol was available for rescue use throughout the study.
- Placebo: Patients received placebo delivered via a single dose dry powder inhaler (SDDPI) once daily (od) in the morning for 3 weeks. Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. The short-acting β2-agonist salbutamol/albuterol was available for rescue use throughout the study.
Arm/Group | Indacaterol 300 μg | Placebo
Number analyzed (Participants) | 78 | 73
Seconds | 586 (30.3) | 475 (31.3)

2. Secondary Outcome: Inspiratory Capacity (IC) Assessed at Rest With Spirometry at the End of Each Treatment Period 60 Minutes Pre-dose
Description: At the end of each 3 week treatment period 60 minutes before inhalation of study drug, IC was measured with spirometry conducted according to internationally accepted standards. The mean of 3 acceptable measurements was calculated and reported in liters.
Time Frame: End of each 3 week treatment period (last day of Weeks 3 and 9)
Population: Modified-intent-to-treat (modified ITT) population: All randomized patients who received at least 1 dose of study drug. The number of patients analyzed for each treatment group was the number with non-missing values for the dependent and independent variables in the mixed model.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Indacaterol 300 μg | Placebo
Number analyzed (Participants) | 78 | 77
Liters | 2.39 (0.034) | 2.25 (0.034)

ADVERSE EVENTS:
Time Frame: Baseline to the end of the study (Week 9)
Description: Adverse events are reported for the safety population which included all patients who received at least one dose of study drug.
Arm/Group | Indacaterol 300 μg | Placebo
Serious Adverse Events (participants affected / at risk) | 3/83 | 1/84
Other Adverse Events (participants affected / at risk) | 6/83 | 10/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Indacaterol 300 μg (N=83) | Placebo (N=84)
Angina pectoris (Cardiac disorders) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Indacaterol 300 μg (N=83) | Placebo (N=84)
Nasopharyngitis (Infections and infestations) | 6 | 6
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.